CLINICAL TRIAL: NCT01427699
Title: A Phase II Study of the Safety, Pharmacokinetics, and Preliminary Efficacy of an Anti-Inflammatory Therapeutic Antibody (MABp1) in Patients With Type 2 Diabetes
Brief Title: A Study of the Safety and Pharmacokinetics of an Anti-Inflammatory Therapeutic Antibody (MABp1) in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-PT011
Record Dates: First submitted 2011-08-31; First posted 2011-09-01 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- T2-18C3 therapeutic antibody (Experimental): 9 subjects will receive the T2-18C3 therapeutic antibody.
  Interventions: Drug: T2-18C3 therapeutic antibody

INTERVENTIONS:
Drug: T2-18C3 therapeutic antibody — 1.25 mg/kg Intravenous infusion every 2 weeks for a total of 4 doses.

SUMMARY:
The purpose of this study is to determine if T2-18C3, a true human monoclonal antibody that blocks inflammation, is safe to use in patients with type 2 diabetes. The study will also be looking at the ability of T2-18C3 to improve control of blood sugar levels in diabetics by blocking inflammation in the pancreas.

DETAILED DESCRIPTION:
This is a phase I, open label study of the safety and pharmacokinetics of T2-18C3 in patients with T2D. Nine patients will receive four biweekly IV infusions of the study drug, T2-18C3, at a dose level of 1.25 mg/kg. These patients will be followed for a total of 90 days to examine safety, pharmacokinetics, and preliminary efficacy.

ELIGIBILITY:
Inclusion Criteria:

* American Diabetes Association (ADA) diagnostic criteria for Type 2 Diabetes (T2D)
* HbA1c >7.0% and ≤ 10%
* Current T2D duration > 3 months at Screening
* T2D and other diseases must be stable. Stable disease is defined as disease which did not require a change in medication or dosing level on 4 or more consecutive days or 7 days in total within 28 days prior to Day 0.
* Age ≥ 18 and ≤ 70 at Screening
* BMI ≥ 23 and ≤ 40 kg/m2
* For female patients of child-bearing age, a negative serum pregnancy test. For patients with reproductive potential, a willingness to utilize adequate contraception (oral contraception plus a mechanical barrier) and not become pregnant (or have their partner[s] become pregnant) during the study
* Agrees not to change diet and exercise regimen during the trial
* Signed and dated Ethics Committee (EC) approved informed consent before any protocol-specific screening procedures are performed

Exclusion Criteria:

* Use of the following medications:

  * Daily use of steroids or aspirin ≥ 700 mg per week
  * Immunosuppressive treatment
  * Thiazolidinediones
  * Concomitant treatment with any other therapeutic antibody, or treatment with any biologic agent that blocks the IL-1 or TNFα signaling pathway
* Change in medication for diabetes within 28 days prior to Day 0, defined as a change in dosing level on 4 or more consecutive days or 7 days in total
* Hemoglobin <10.0 g/dL, WBC <3.0 x 103/mm3 , platelet count <125 x 103/mm3, creatinine > 1.5mg/dL, AST/ALT >2 x ULN, alkaline phosphatase >2 x ULN
* Abnormal, untreated T3, T4, thyroglobulin, or TSH levels or history of Grave's disease
* Known HIV antibody, hepatitis B surface antigen and/or hepatitis C antibody
* History of malignancy within 5 years prior to study entry other than carcinoma in situ of the cervix, or adequately treated, nonmetastatic squamous or basal cell carcinoma of the skin
* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies
* History of tuberculosis, positive PPD test, active atopic disease requiring medication, or asthma
* Infectious disease:

  * CRP >30 mg/L, fever, or infection requiring treatment with antibiotics within 3 weeks prior to Screening
  * History of recurrent infection or predisposition to infection
  * Active leg or foot ulcer
* Immunodeficiency
* Female patients who are pregnant, planning to become pregnant during the course of the study, or breast-feeding
* Receipt of a live (attenuated) vaccine within 3 months prior to Screening
* Major surgery within 28 days prior to Day 0
* Participation in an investigational drug or device trial within 30 days prior to Screening

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2011-06-30 (Actual); Primary Completion 2012-10-31 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability | 90 days
  The safety and tolerability of T2-18C3 will be determined by observing patients for clinical adverse events, changes in vital signs, and changes in laboratory parameters such as hematology and chemistry.

SECONDARY OUTCOMES:
Pharmacokinetics | 90 days
  Serum levels of T2-18C3 will be measured in patients
Preliminary Efficacy | 90 days
  The ability of T2-18C3 to improve glycemic control will be measured by comparing the change in glycosylated hemoglobin levels of patients from baseline to day 90.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Basel, Basel, Switzerland

REFERENCES:
- [Derived] Timper K, Seelig E, Tsakiris DA, Donath MY. Safety, pharmacokinetics, and preliminary efficacy of a specific anti-IL-1alpha therapeutic antibody (MABp1) in patients with type 2 diabetes mellitus. J Diabetes Complications. 2015 Sep-Oct;29(7):955-60. doi: 10.1016/j.jdiacomp.2015.05.019. Epub 2015 Jun 3. PMID 26139558